CLINICAL TRIAL: NCT05914779
Title: Impact of Early Antibiotics on Non-Traumatic Out of Hospital Cardiac Arrest (OHCA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Adeel Ajwad Butt, Senior Consultant in Infectious Diseases, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRGC-05-SI-18-356
Record Dates: First submitted 2023-05-30; First posted 2023-06-22 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Infection, Bacterial; Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Bacterial Infections; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subject with antibiotics treatment (Experimental): Individuals with low risk of infection after OHCA will be randomized to either 1) early antibiotics, or 2) no antibiotics.
  Experimental arm received antibiotics as per local hospital clinical care pathways and physician choice.
  Interventions: Other: with antibiotics treatment
- Subjects with no antibiotics treatment (Active Comparator): Individuals with low risk of infection after OHCA will be randomized to either 1) early antibiotics, or 2) no antibiotics.
  Active comparator arm will receive no antibiotics,
  Interventions: Other: No use of antibiotics

INTERVENTIONS:
Other: No use of antibiotics — Subjects will be randomized into antibiotics and no antibiotics groups based on inclusion and exclusion criteria
  Arms: Subjects with no antibiotics treatment
Other: with antibiotics treatment — with antibiotics treatment
  Arms: Subject with antibiotics treatment

SUMMARY:
Specific Aim : The specific aim is to conduct a randomized prospective clinical trial to determine whether no antibiotics in OHCA patients in the ED with very low likelihood of infection is non-inferior to early antibiotic treatment. Hypothesis a: 28-day all-cause mortality will be non-inferior in OHCA patients with very low likelihood of infection who do not receive antibiotic therapy compared with those who receive early antibiotic therapy Hypothesis b: There will be no difference in subsequent incidence of proven infections in the no antibiotics vs, early antibiotics groups Hypothesis c: There will be no difference in the length of ICU stay and overall hospital stay in the early antibiotics vs. no antibiotics groups

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* ● Adults aged >18 years, presenting to HGH ED after out-of-hospital cardiac arrest

  * Patients with low likelihood of infection as per the definitions provided above
  * Ability to obtain informed consent from the subjects or their next of kin/family member/legal surrogate in case of incapacitation due to sedation, mechanical ventilation, etc. In case the next of kin is not available, an independent physician who is not a part of the investigative team will complete and sign the checklist as per HMC Policy "RES 11026_Appendix 6.5". (see section 4.1.3 for details) A member of the investigative team and a witness will also sign this form before the potential subject is enrolled in the study.

Exclusion Criteria:

* Patients who have clear evidence of infection, as defined by criteria for the study.

  * Patients who have received antibiotics within the last 1 week prior to admission.
  * Patients with malignancy, except those who have been cured or in complete remission.
  * Females with known pregnancy.
  * Known immunocompromised states (including HIV/AIDS, transplant recipients on immunosuppressant drugs, long-term [> 3 weeks of prednisone >5mg/day equivalent] steroid therapy).
  * Patients on immunologic disease modifying agents (commonly known as "biologics")
  * Patients considered "brain-dead" or "vegetative state"
  * Patients transferred from another hospital, long term care facility or institution
  * Neutropenia (total WBC <1,500/mm3 or absolute neutrophil count of <1,000/mm3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality. likelihood of infection whether they receive early antibiotic therapy or not. | 28-day
  Primary outcome measure is 28-day all-cause mortality in persons who receive no antibiotics compared with those who receive early antibiotics in OHCA patients.

CONTACTS AND LOCATIONS:
Overall Officials: Adeel A Butt, MBBS, MS, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Baladīyat ad Dawḩah, Qatar

IPD SHARING:
Plan to Share IPD: No